CLINICAL TRIAL: NCT03281772
Title: Technology Assisted Management of Uncontrolled Hypertension (TEAM-HTN): a Pilot Study
Brief Title: Uncontrolled Hypertension Management (TEAM-HTN)
Acronym: TEAM-HTN
Status: Terminated | Type: Observational
Why Stopped: PI retired before recruitment was started.
Sponsor: Madigan Army Medical Center (U.S. Federal Agency)
Collaborators: Telemedicine & Advanced Technology Research Center (Other); Analytics4Medicine, LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: AAMTI 6422
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Uncontrolled Hypertension
Keywords: hypertension; clinical decision support software; renin; aldosterone
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Provider: Consented providers with prescriptive privileges will use the clinical decision software - provider portal to manage study patients with uncontrolled hypertension for 6 months. Participants will conduct a baseline face-to-face visit with study patients, access the program daily to check for patient high blood pressure alerts and lab results, conduct virtual visits as needed every 7 - 10 days, track the time and number of patients managed using the program and complete two questionnaires.
  Interventions: Other: Clinical Decision Software - provider portal
- Patients Phase 1: All consented participants provider or self-referred with uncontrolled HTN, completed a demographic questionnaire and received instruction on proper technique for checking home BPs using a study-provided, digital BP monitor with an appropriate-sized arm cuff. Readings were taken three days per week at a consistent time of day of their choosing between 8 AM and noon and 4PM and 8 PM (morning surge and chronotherapy trough). Baseline readings, the first 10 home readings taken over 10 days, were used to determine phase 2 eligibility. If 4 or more baseline readings were above recommended individualized JNC 8 BP goals set by their primary care provider, patients met criteria for rHTN and advanced to phase 2. Phase 1 patients advancing to phase 2 (met criteria for rHTN) acted as their own controls. Patients were not screened for secondary causes of HTN prior to entering phase 2.
  Interventions: Other: Clinical Decision Software - patient portal
- Patients Phase 2: Phase 2 patients continued checking BPs as in phase 1, had morning renin and aldosterone levels drawn while on their current medications, and were systematically screened by study providers for secondary causes of HTN using the CDST's diagnostic matrix. If aldosterone was significantly elevated (> 20 ng/dl) and/or the aldosterone/renin ratio (ARR) was over 25, a 3-week drug wash out interval and repeat labs were recommended in the matrix for the work up of primary aldosteronism (PA). Due to institutional review board (IRB) stipulations, the actual workup for PA or other secondary causes of rHTN was managed by patients' PCP. Electrolytes were drawn as clinically indicated.
  Interventions: Other: Clinical Decision Software - patient portal

INTERVENTIONS:
Other: Clinical Decision Software - provider portal — As noted in Arms
  Groups: Provider
Other: Clinical Decision Software - patient portal — As noted in Arms
  Groups: Patients Phase 1; Patients Phase 2

SUMMARY:
Current guideline directed medical therapies (GDMT) for hypertension (HTN) endorse a trial and error approach based on drug class. This pilot study will evaluate the efficacy of a Clinical Decision Support (CDS) program to assist providers with delivering a more personalized approach using individual renin-aldosterone levels and the mechanism of action of medications included in GDMT recommendations. The overarching goal is to achieve HTN control rates above the 2014 National Health and Nutrition Examination Survey reported rate of 53% in a timely fashion, by individualizing medication management, thereby reducing the patient risk of stroke, heart and renal disease, and other devastating HTN-related outcomes.

DETAILED DESCRIPTION:
Current guideline directed medical therapies (GDMT) for hypertension (HTN) endorse a trial and error approach based on drug class. This pilot study will evaluate the efficacy of a Clinical Decision Support (CDS) program to assist providers with delivering a more personalized approach using individual renin-aldosterone levels and the mechanism of action of medications included in GDMT recommendations. Current research suggests underlying mechanisms of HTN can be categorized by renin and aldosterone levels into approximately 50 categories and sub-categories. Timely identification of a patients' category is challenging for clinicians and possibly a contributing factor to the low rates of HTN control reported in the 2014 National Health and Nutrition Examination Survey (NHANES) of 53%. The overarching goal of this study is to achieve HTN control rates above the 2014 NANES rate in a timely, cost-effective manner by individualizing medication management, thereby reducing the patient risk of stroke, heart and renal disease, and other devastating HTN-related outcomes. Specific aims are: 1) evaluate the efficacy of the CDS software program to assist providers in identifying and matching the underlying mechanisms of HTN with the mechanism of action of antihypertensive medications to achieve better HTN control rates than the 53% reported in the 2014 NHANES data, 2) assess the efficacy of the CDS program across prescribing provider levels (MD/DO, residents, and APRN/PA), and 3) Determine the impact of the CDS program on: a) medication costs, b) provider management time, c), provider and patient satisfaction with and perception of usability and efficacy of the CDS program to manage their blood pressure. This 2-phase, prospective, within-subjects, repeated measures pilot study will enroll up to 20 multi-level providers with prescriptive authority and 160 military beneficiaries with uncontrolled HTN in the Northwest to evaluate the efficacy, feasibility, and usability of a CDS program to improve blood pressure control over a six-month period.

ELIGIBILITY:
Inclusion Criteria:

1. Providers with prescriptive authority practicing in outpatient clinics at a military treatment facility in the Northwest.
2. Patients 18 years or older with uncontrolled hypertension receiving care in an outpatient setting that can give a valid consent (over age 18 years, the ability to read and understand English, and cognitively intact). Active duty service members who will not be deployed or due to change duty station for the duration of the study.

   -

   Exclusion Criteria:

1. Credentialed providers without prescribing privileges in good standing. 2. Age less than 18 years, night shift workers, anyone who cannot give a valid informed consent, pregnant or breast feeding women, prisoners, patients on renal dialysis, transplant recipients, life expectancy less than 1 year, and those disqualified during screening procedures.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Credentialed providers with prescriptive authority and patients with uncontrolled hypertension practicing at or enrolled in a military treatment facility in the Pacific Northwest.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2017-01-24 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Patients with controlled hypertension | 6 months
  Percent of systolic and diastolic blood pressure readings within patient-specific target goals averaged in 10-day cycles at least 70% of the time.

SECONDARY OUTCOMES:
Provider Satisfaction | 6 months
  Provider satisfaction with efficacy, feasibility and usability of the clinical decision software program
Patient Satisfaction | 6 months
  Patient satisfaction with efficacy, feasibility and usability of the clinical decision software program
Provider time | 6 months
  Time in minutes each provider spends per patient managing uncontrolled hypertension.
Medication costs | 6 months
  Costs of medications per patient to achieve controlled hypertension using a published relative value scale
Time to reach blood pressure goals | 6 months
  Number of days from enrollment patients are not at target (70% control rate)
Patients with controlled hypertension by provider | 6 months
  Number of patients per provider level (MD, DO, Nurse Practitioner, Physician Assistant) with controlled hypertension

CONTACTS AND LOCATIONS:
Overall Officials: Leilani A. Siaki, PhD, Principal Investigator — Madigan Army Medical Center
Locations (1):
- Madigan Army Medical Center, Tacoma, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] James PA, Oparil S, Carter BL, Cushman WC, Dennison-Himmelfarb C, Handler J, Lackland DT, LeFevre ML, MacKenzie TD, Ogedegbe O, Smith SC Jr, Svetkey LP, Taler SJ, Townsend RR, Wright JT Jr, Narva AS, Ortiz E. 2014 evidence-based guideline for the management of high blood pressure in adults: report from the panel members appointed to the Eighth Joint National Committee (JNC 8). JAMA. 2014 Feb 5;311(5):507-20. doi: 10.1001/jama.2013.284427. PMID 24352797
- [Background] Kisaka T, Ozono R, Ishida T, Higashi Y, Oshima T, Kihara Y. Association of elevated plasma aldosterone-to-renin ratio with future cardiovascular events in patients with essential hypertension. J Hypertens. 2012 Dec;30(12):2322-30. doi: 10.1097/HJH.0b013e328359862d. PMID 23107914
- [Background] Weber MA, Schiffrin EL, White WB, Mann S, Lindholm LH, Kenerson JG, Flack JM, Carter BL, Materson BJ, Ram CV, Cohen DL, Cadet JC, Jean-Charles RR, Taler S, Kountz D, Townsend R, Chalmers J, Ramirez AJ, Bakris GL, Wang J, Schutte AE, Bisognano JD, Touyz RM, Sica D, Harrap SB. Clinical practice guidelines for the management of hypertension in the community a statement by the American Society of Hypertension and the International Society of Hypertension. J Hypertens. 2014 Jan;32(1):3-15. doi: 10.1097/HJH.0000000000000065. No abstract available. PMID 24270181
- [Background] Moran AE, Odden MC, Thanataveerat A, Tzong KY, Rasmussen PW, Guzman D, Williams L, Bibbins-Domingo K, Coxson PG, Goldman L. Cost-effectiveness of hypertension therapy according to 2014 guidelines. N Engl J Med. 2015 Jan 29;372(5):447-55. doi: 10.1056/NEJMsa1406751. PMID 25629742
- [Background] SPRINT Research Group; Wright JT Jr, Williamson JD, Whelton PK, Snyder JK, Sink KM, Rocco MV, Reboussin DM, Rahman M, Oparil S, Lewis CE, Kimmel PL, Johnson KC, Goff DC Jr, Fine LJ, Cutler JA, Cushman WC, Cheung AK, Ambrosius WT. A Randomized Trial of Intensive versus Standard Blood-Pressure Control. N Engl J Med. 2015 Nov 26;373(22):2103-16. doi: 10.1056/NEJMoa1511939. Epub 2015 Nov 9. PMID 26551272
- [Background] Yoon SS, Fryar CD, Carroll MD. Hypertension prevalence and control among adults: United States, 2011-2014. Data from the National Health and Nutrition Examination Survey. http://www.cdc.gov/nchs/products/databriefs/db220.htm . Accessed March 18, 2016.
- [Background] Bochud M, Burnier M, Guessous I. Top Three Pharmacogenomics and Personalized Medicine Applications at the Nexus of Renal Pathophysiology and Cardiovascular Medicine. Curr Pharmacogenomics Person Med. 2011 Dec;9(4):299-322. doi: 10.2174/187569211798377135. PMID 23049672
- [Background] Rosendorff C, Lackland DT, Allison M, Aronow WS, Black HR, Blumenthal RS, Cannon CP, de Lemos JA, Elliott WJ, Findeiss L, Gersh BJ, Gore JM, Levy D, Long JB, O'Connor CM, O'Gara PT, Ogedegbe G, Oparil S, White WB; American Heart Association, American College of Cardiology, and American Society of Hypertension. Treatment of hypertension in patients with coronary artery disease: a scientific statement from the American Heart Association, American College of Cardiology, and American Society of Hypertension. Hypertension. 2015 Jun;65(6):1372-407. doi: 10.1161/HYP.0000000000000018. Epub 2015 Mar 31. No abstract available. PMID 25828847
- [Background] Deal, P. (2011). Hypertension: More Soldiers die from silent killer than combat. Army News Front Page. Retrieved October 24, 2015 from: http://www.army.mil/article/59005/
- [Background] Wang G, Fang J, Ayala C. Hypertension-associated hospitalizations and costs in the United States, 1979-2006. Blood Press. 2014 Apr;23(2):126-33. doi: 10.3109/08037051.2013.814751. Epub 2013 Jul 25. PMID 23885763